CLINICAL TRIAL: NCT06319443
Title: Daily Vinegar Ingestion and 24-Hour Blood Glucose Control in Adults With Glucose Intolerance: A Randomized Crossover Trial
Brief Title: Daily Vinegar Ingestion and 24-Hour Blood Glucose Control
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Arizona State University (Other)
Responsible Party: Principal Investigator, Carol Johnston, Professor and Associate Dean, Arizona State University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: STUDY00019235
Record Dates: First submitted 2024-03-13; First posted 2024-03-20 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Glucose Intolerance
Keywords: glucose; continuous glucose monitoring; vinegar
MeSH Terms: conditions — Glucose Intolerance | interventions — Acetic Acid

STUDY DESIGN:
Intervention Model Description: This is a 9-day trial. Participants will be fitted with a continuous glucose monitor and follow their typical diet and activity patterns. Participants will be randomized to ingest 2 tablespoons of vinegar twice daily (diluted in water) or a vinegar pill for the first 4 days on the trial. On day 5 of the trial participants will consume the alternate treatment for trial days 5-8. Dietary intake will be recorded daily using a fitness app. Physical activity will be assessed at baseline and on study day 4 and 8. On day 9, participants will return to the test site for device removal.
Who Masked: Participant
Masking Description: Liquid and pill vinegar will be the treatments. The pill is the 'control' as the level of acetic acid is below the amount needed for an antiglycemic effect (a fact not realized by the participant).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Liquid vinegar (Experimental): Liquid vinegar (6% acidity) consumed at a dosage of 2 tablespoons (diluted in water and consumed at mealtime) twice daily (4 tablespoons total per day).
  Interventions: Dietary Supplement: Liquid vinegar
- Vinegar pill (Placebo Comparator): One pill consumed daily in the morning.
  Interventions: Dietary Supplement: vinegar pill

INTERVENTIONS:
Dietary Supplement: Liquid vinegar — 3.5 g acetic acid
  Arms: Liquid vinegar
Dietary Supplement: vinegar pill — 0.022 g acetic acid
  Arms: Vinegar pill

SUMMARY:
When linking dietary interventions and blood glucose management, much of the existing research - particularly studies exploring the effects of vinegar - has relied on discrete readings from the conventional testing methods: blood samples or glucometers. These methods lack the capacity to provide insights into blood glucose dynamics 24/7.

Recognizing this gap, the current study aims to utilize continuous glucose monitoring to examine the impact of daily vinegar ingestion on glucose variability in adults identified as glucose intolerant.

DETAILED DESCRIPTION:
Participants are randomly assigned to either Group A or Group B using the Microsoft Excel randomization function. Group A will be instructed to consume 4 tablespoons of red wine vinegar (2 tablespoons diluted in water at the start of the lunch and the dinner meals) for the first 4 days of the trial. Conversely, participants in Group B will ingest the placebo for the initial 4 days, ingesting one pill daily upon waking in the morning. On days 5-9, participants will switch to the opposite treatment. The red wine vinegar dosage (4 tablespoons containing 3.5 g acetic acid - this is the amount of acetic acid in a large 4-inch dill pickle), and the placebo vinegar pill dosage (one pill containing 0.022 g acetic acid) will be taken daily during the trial. On visit 1, anthropometric measurements, including height, weight, and body composition (lean fat mass and body fat mass), will be measured, and the continuous glucose monitor will be placed on the upper arm. The participants will be instructed to fast >8 hours (no food or beverages with the exception of water) ahead of visit 1. To ensure accurate use and data collection, researchers discussed the operation of CGM devices and that these waterproof devices are to be continuously worn during the entire 9-day trial and will be removed on day 9 (visit 2).

ELIGIBILITY:
Inclusion Criteria:

* glucose intolerance (defined as one of the following: fasting glucose >99 mg/dl; diagnosis of prediabetes or diabetes; history of gestational diabetes)
* 18 years of age or older
* sedentary or moderately active (defined as a score ≤ 24 on the Godin-Shepard Leisure Time Physical Activity Questionnaire)

Exclusion Criteria:

* currently adhering to a non-typical diet that would impact carbohydrate intake (including weight loss diets)
* medication/drug use that has not been consistent for the previous 3 months or will be discontinued during the trial
* any acute illness
* regular smokers, pregnant or lactating women, or individuals taking insulin
* Unwilling to tolerate vinegar ingestion

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2024-03-26 (Actual); Primary Completion 2024-12-15 (Actual); Study Completion 2025-07-15 (Actual)

PRIMARY OUTCOMES:
Average glucose | Four days
  The average blood glucose concentration for each 4-day period
Glucose: time in range | Four days
  The average time over 4 days that blood glucose falls in the reference range

CONTACTS AND LOCATIONS:
Locations (1):
- 850 PBC, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No